CLINICAL TRIAL: NCT06998667
Title: Cooling Solutions for Outdoor Workers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shuchi Anand, Associate Professor in Nephrology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 80246
Record Dates: First submitted 2025-05-20; First posted 2025-05-31 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hyperthermia; Heat Acclimation and Thermotolerance
Keywords: outdoor work; heat stress; kidney injury; cooling interventions
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Heat Illness Prevention (Active Comparator): Standard CAL-OSHA workplace heat illness prevention interventions, which require availability of cool, potable water; availability of shade when temperatures exceed 80F; and encouragement of rest for cool down breaks.
  Interventions: Behavioral: Standard Heat Illness Prevention Measures
- Cooling bandana with Standard Heat Illness Prevention Measures (Experimental): Provision of a bandana with slow-evaporation polymer for use during work, in addition to standard CAL-OSHA workplace heat illness prevention interventions
  Interventions: Behavioral: Standard Heat Illness Prevention Measures; Other: Cooling bandana
- Cooling glove with standard Heat Illness Prevention (Experimental): Provision of a glove with ability to circulate cool water, for use during breaks, in addition to standard CAL-OSHA workplace heat illness prevention interventions
  Interventions: Behavioral: Standard Heat Illness Prevention Measures; Other: Cooling glove

INTERVENTIONS:
Behavioral: Standard Heat Illness Prevention Measures — Standard CAL-OSHA workplace heat illness prevention interventions, which require availability of cool, potable water; availability of shade when temperatures exceed 80F; and encouragement of rest for cool down breaks
Other: Cooling bandana — Cooling bandana embedded with a polymer to slow evaporation
  Arms: Cooling bandana with Standard Heat Illness Prevention Measures
Other: Cooling glove — Cooling glove with ability to circulate cool water interface with palmar skin
  Arms: Cooling glove with standard Heat Illness Prevention

SUMMARY:
The investigators aim to test the effectiveness of two cooling interventions in reducing the core temperature of outdoor workers.

DETAILED DESCRIPTION:
Workers in a variety of US industries-construction workers, welders, farmers, firefighters, and warehouse workers among them-are at risk for hyperthermia during work, yet very few interventions are being developed to mitigate heat related organ injury, particularly when workers do not have obvious symptoms of heat related illness. The investigators plan to test whether two active cooling technologies can help mitigate hyperthermia and risk for kidney injury. This work will enhance worker safety using evidence-based technology.

To accomplish the aims of testing two active cooling interventions, the investigators plan to implement a case-cross over randomized control trial design at the work site conducted in partnership with an employer and with 30 workers at risk for hyperthermia. Over three sequential weeks, the investigators will measure rate of core temperature change (primary outcome). Secondary outcomes will include changes in kidney injury markers; changes in worker productivity; and worker acceptability of interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Anticipated to be working in the same job category for the duration of the study
3. Able to communicate in English or Spanish

Exclusion Criteria:

1. Cannot provide informed consent
2. Weight less than 40 kg
3. Inability to swallow pills
4. Known history of having a pacemaker or ICD
5. Pregnancy as determined by self report and confirmed on Day 1
6. Gastrointestinal disorders (e.g., gastroparesis, prior surgery on GI tract with the exception of appendectomy or cholecystectomy, diverticulosis or inflammatory bowel disease)
7. Plan for an elective MRI in the 7 days post last planned pill ingestion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Core Temperature | up to 10 hours
  Rate of core temperature change as measured by core temperature pill

CONTACTS AND LOCATIONS:
Overall Officials: Shuchi Anand, MD, Principal Investigator — Stanford University; Julie Parsonnet, MD, Principal Investigator — Stanford University; Maria Montez Rath, mrath@stanford.edu, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
At the moment we plan to reserve individual participant data for current project only